CLINICAL TRIAL: NCT07037875
Title: A Randomized, Phase 3, Double-blind, Double-dummy, Active Comparator-controlled Multicenter Study to Evaluate the Efficacy and Safety of 2 Doses of Linaprazan Glurate Compared to Lansoprazole in 4 or 8 Weeks Healing in Participants With Erosive Esophagitis (EE) Due to Gastroesophageal Reflux Disease (GERD) of Los Angeles (LA) Grades A to D
Brief Title: A Study Comparing the Effect and Safety of Linaprazan Glurate to Lansoprazole in Participants With Erosive Esophagitis (EE) Due to Gastroesophageal Reflux Disease (GERD)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cinclus Pharma Holding AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX842A2301; 2024-518714-31-00 (EU CTIS Number); UTN U1111-1315-2237 (Other: World Health Organization)
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — BID protein, human; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Linaprazan glurate 50 mg BID (Experimental)
  Interventions: Drug: Linaprazan glurate 50 mg Twice Daily (BID)
- Group 2: Linaprazan glurate 50 mg QD (Experimental)
  Interventions: Drug: Linaprazan Glurate 50 mg Once Daily (QD)
- Group 3: Lansoprazole 30 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole 30 mg Once Daily (QD)

INTERVENTIONS:
Drug: Linaprazan glurate 50 mg Twice Daily (BID) — Participants in this group will receive a total daily dose of 100 mg of linaprazan glurate, administered as 50 mg in the morning and 50 mg in the evening.
  In the morning, they take one 50 mg linaprazan glurate tablet along with a placebo capsule that matches the appearance of the lansoprazole capsule. In the evening, they take another 50 mg linaprazan glurate tablet, without any additional placebo.
  Arms: Group 1: Linaprazan glurate 50 mg BID
Drug: Linaprazan Glurate 50 mg Once Daily (QD) — Participants in this group will receive a total daily dose of 50 mg of linaprazan glurate, taken once daily in the morning.
  In the morning, they take one 50 mg linaprazan glurate tablet along with a placebo capsule that mimics the lansoprazole capsule. In the evening, they take a placebo tablet that mimics the appearance of the linaprazan glurate tablet.
  Arms: Group 2: Linaprazan glurate 50 mg QD
Drug: Lansoprazole 30 mg Once Daily (QD) — Participants in this group will receive a total daily dose of 30 mg of lansoprazole, taken once daily in the morning.
  In the morning, they take one 30 mg lansoprazole capsule along with a placebo tablet that mimics the linaprazan glurate tablet. In the evening, they take another placebo tablet resembling linaprazan glurate.
  Arms: Group 3: Lansoprazole 30 mg QD

SUMMARY:
The goal of this clinical trial is to find out how well linaprazan glurate can heal erosive esophagitis (EE) caused by gastroesophageal reflux disease (GERD), compared to lansoprazole, a commonly used medication. Researchers will also evaluate whether linaprazan glurate:

* Reduces heartburn symptoms more effectively than lansoprazole
* Is safe and well tolerated, based on physical exams, blood tests, and vital signs (heart rate, blood pressure, temperature, and breathing rate)
* Causes any side effects during treatment
* Has different effects depending on how much of the drug is in the blood
* Works differently depending on participants' genes

Participants must be between 18 to 80 years old and have EE due to GERD confirmed by an endoscopy. Participants cannot join if they have an active Helicobacter pylori (HP) infection or were treated for HP in the past 6 weeks or have taken antibiotics or bismuth-containing drugs in the past 6 weeks.

The study is a randomized, double-blind, active comparator-controlled trial lasting up to 4 months. Randomized means that participants are assigned by chance (like flipping a coin) to one of the treatment groups and double-blind means neither the participants nor the study team will know which treatment is given. Participants will be placed into one of three groups (about 167 people in each group):

* Linaprazan glurate 50 mg twice a day
* Linaprazan glurate 50 mg once a day
* Lansoprazole 30 mg once a day

Everyone will take 2 tablets and 1 capsule by mouth daily for 8 weeks. Some tablets or capsules will be placebos (look like medicine but contain no active drug). Participants will:

* Undergo an endoscopy in the beginning and after 4 weeks of treatment
* If healing is not observed, another endoscopy may be done at 8 weeks
* During the procedure, doctors will use a thin, flexible tube with a camera to look at the esophagus and take small tissue samples (biopsies)
* Have blood and urine tests at clinic visits to check overall health
* Receive electrocardiograms (ECGs) to monitor heart function
* Complete daily questionnaires on an electronic device about symptoms and experiences

ELIGIBILITY:
Inclusion Criteria:

1. The participant understands and voluntarily signs an Informed Consent Form (ICF) prior to initiation of any study-related assessments/procedures.
2. Male or female participants aged 18 to 80 years, inclusive, at the time of signing the ICF.
3. The participant is willing and able to comply with all aspects of the protocol (including endoscopies, PK sampling, tablet and capsule swallowing, electronic device [e-device] completion, etc.).
4. The participant has endoscopically confirmed EE due to GERD of LA grades A to D during the Screening Period as assessed in Central Review by an Independent Review Committee (IRC).

Exclusion Criteria:

1. Ongoing infection with HP or diagnosis and treatment of HP infection within 6 weeks of randomization OR any treatment with antibiotics or bismuth containing drugs within 6 weeks of randomization.
2. History or presence of any clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, neurological disease or disorder, or psychiatric diagnosis which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the study results or the participant's ability to participate in the study. The following examples are conditions that would exclude the patient from participating:

   1. History of myocardial infarction/acute coronary syndrome within 3 months prior to Screening.
   2. History of ventricular arrhythmia or implanted cardioverter defibrillator.
   3. Symptomatic congestive heart failure (New York Heart Association class 3-4).
   4. Family history of/diagnosis of hereditary arrhythmia syndrome.
   5. History of adult asthma that required intensive treatment in an emergency room.
3. History of malignancy of any organ system (other than completely treated localized basal cell carcinoma or non-metastatic squamous cell carcinoma of the skin or in situ cervical carcinoma), within the past 5 years.
4. Solitary esophageal ulcer in the proximal two-thirds of the esophagus, untreated Barrett's esophagus or any other condition affecting the esophagus, including eosinophilic esophagitis; esophageal varices; viral or fungal infection; esophageal stricture*; a history of radiation therapy, radiofrequency ablation, endoscopic mucosal resection, or cryotherapy to the esophagus; or any history of caustic or physiochemical trauma.

   *Note: Patients with diagnosis of Schatzki's ring (mucosal tissue ring around lower esophageal sphincter) are eligible to participate, unless history of dilatation within 3 months of Screening.
5. History of any surgical or medical condition which might significantly alter the GERD status or the absorption, distribution, metabolism, or excretion of drugs. The Investigator is to be guided by evidence of any of the following: history of major GI surgery such as gastrectomy, gastroenterostomy, any bariatric surgery, bowel resection, or transjugular intrahepatic portosystemic shunt. Nissen fundoplication is not exclusionary as long as the patient is eligible according to other criteria.
6. Known severe atrophic gastritis as assessed from medical history or upper endoscopy during Screening.
7. Zollinger-Ellison syndrome or other gastric acid hypersecretory conditions.
8. History of treatment course with lansoprazole within 2 months prior to Screening.
9. Current peptic ulcer.
10. Body mass index (BMI) ≤ 18 and ≥ 40 kg/m² at Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Healing of EE at Week 4 as assessed by endoscopy in participants with Baseline EE LA grades C/D. | From enrollment to the end of treatment at 4 weeks.

CONTACTS AND LOCATIONS:
Locations (75):
- Bulgaria (15):
  - Medical Center "Orange", Sofia, Sofia City Province
  - Multiprofile Hospital for Active Treatment - "Vita", Sofia, Sofia City Province
  - Diagnostic and Consulting Center Alexandrovska, Sofia, Sofia City Province
  - Diagnostic Consultative Center - Focus-5, Sofia, Sofia City Province
  - Medical Center Hera, Sofia, Sofia City Province
  - University Multiprofile Hospital for Active Treatment "Tsaritsa Yoanna - ISUL", Sofia, Sofia City Province
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov, Sofia, Sofia City Province
  - 20th Diagnostic Consultancy Center, Sofia, Sofia City Province
  - Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski - 2003" OOD, Dupnitsa
  - Multiprofile Hospital For Active Treatment St. Ivan Rilski Gorna Oriahovitsa EOOD, Gorna Oryahovitsa
  - Medical Center Hera, Kyustendil
  - University Multiprofile Hospital for Active Treatment "Sveta Marina", Pleven
  - Multiprofile Hospital for Active Treatment "Sveti Panteleymon", Plovdiv
  - Diagnosis - Consulting Centre 1, Sliven
  - First Private Hospital Vratsa, Vratsa
- Czechia (7):
  - SurGal Clinic s.r.o., Brno
  - Military Hospital Brno, Internal Department, Brno
  - University Hospital Brno, Brno
  - PreventaMed s.r.o., Olomouc
  - Gastromedic s.r.o., Pardubice
  - Hospital Prachatice a.s., Prachatice
  - Endohope Morava s.r.o., Zábřeh
- Georgia (11):
  - Khozrevanidze's Clinic, Batumi
  - JSC Georgian Clinics, Kutaisi
  - LTD Aversi Clinic, Marneuli
  - LTD Krol Medical Corporation, Tbilisi
  - The New Hospitals, Tbilisi
  - Israeli - Georgian Medical Research Clinic Healthycore LLC, Tbilisi
  - Janmrtelobis Sakhli LLC, Tbilisi
  - LLC Geo Hospitals, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LEPL The First University Clinic of Tbilisi State Medical University, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LLC, Tbilisi
- Germany (3):
  - Diakonie Hospital, Mannheim, Baden-Wurttemberg
  - Medical Care Unit Dachau, Dachau, Bavaria
  - Clinic for Internal Medicine Munich-Sued, Munich, Bavaria
- Hungary (11):
  - Bekes County Central Hospital Dr. Rethy Pal Member Hospital, 4th Department of Internal Medicine - Gastroenterology - Hepatology, Békéscsaba
  - G1 Institute, Budapest
  - Clinexpert Ltd. Budapest, Budapest
  - Obuda Healthcare Center Ltd., Budapest
  - Synexus Hungary Ltd., Budapest
  - Central Hospital of Northern Pest - Military Hospital, Department of Gastroenterology, Budapest
  - Main Railway Outpatient Clinic Debrecen, Department of Gastroenterology, Debrecen
  - Heves County Markhot Ferenc Teaching Hospital and Clinic, Department of General and Vascular Surgery, Eger
  - University of Szeged, Department of Internal Medicine- Western Site, Szeged
  - Fejer County St. Gyorgy University Teaching Hospital, Department of Internal Medicine I, Székesfehérvár
  - Javorszky Odon Hospital Vac, Department of Gastroenterology, Vác
- Poland (25):
  - NZOZ Specialist Gastrology Centre GASTROMED, Bialystok
  - "MEDIS" Medical Center, Bydgoszcz
  - NZOZ KERmed Medical Centre, Bydgoszcz
  - CLINSANTE Clinical Research Centre Ewa Galczak-Nowak, Malgorzata Trzaska, Bydgoszcz
  - St. John Paul 2nd Municipal Hospital in Elblag, Department of Internal Diseases, Elblag
  - Synexus Polska Sp. z o.o. Branch in Gdansk, Gdansk
  - Synexus Polska Sp. z o.o. Branch in Katowice, Katowice
  - "Vita Longa" Non-Public Healthcare Facility, Limited Liability Company, Katowice
  - Independent Public Healthcare Facility University Hospital in Krakow, NSSU Endoscopy Department, Krakow
  - FutureMeds Krakow, Krakow
  - Independent Public Healthcare Facility, Norbert Barlicki University Teaching Hospital No. 1 of the Medical University in Lodz, Clinical Department of General Gastroenterology and Oncology, Lodz
  - Hospital of Brothers Hospitallers of Saint John of God In Lodz, Endoscopy Lab, Lodz
  - Oswiecim Clinical Trial Centre, Oświęcim
  - EMC Medical Institute Joint Stock Company, CERTUS Private Healthcare Facility Hospital No. 1, CERTUS Private Healthcare Facility Ambulatories, Poznan
  - Synexus Polska Sp. z o.o. Branch in Poznan, Poznan
  - New health-CK, Kieltucki and partners g.p., Staszów
  - Gastromed Sp. z o.o. (LLC), Torun
  - FutureMeds Warsaw Center, Warsaw
  - Therapia Nova, Warsaw
  - ETG Warszawa, Warsaw
  - Futuremeds Targowek, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Medical Centre Oporow, Wroclaw
  - FutureMeds Wroclaw, Wroclaw
  - ETG Zamosc, Zamość
- Romania (3):
  - Colentina Clinical Hospital, Department of Gastroenterology, Bucharest
  - Cluj Napoca County Emergency Clinical Hospital, Internal Medicine III, Cluj-Napoca
  - TVM MED SERV SRL, Medical Center for Gastroenterology, Hepatology and Digestive Endoscopy, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: No